CLINICAL TRIAL: NCT06908005
Title: Development and Prognostic Validation of RaFIST: A Radiomics-Based Tool for Intratumoral Fibrosis Stratification in Non-Small Cell Lung Cancer
Brief Title: RaFIST: A Radiomics-Based Tool for Intratumoral Fibrosis Stratification in Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Guangming Lu, Professor, Jinling Hospital, China
Other Study IDs: 2025-DZLC-02
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer - Non Small Cell
Keywords: NSCLC; radiomics; PFS; fibrosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- training set
  Interventions: Other: CT radiomic analysis; Other: Fibrosis assessment
- external test set
  Interventions: Other: CT radiomic analysis; Other: Fibrosis assessment

INTERVENTIONS:
Other: CT radiomic analysis — Radiomic features of tumor tissue
Other: Fibrosis assessment — Fibrosis quantification was performed on picrosirius red (PSR)-stained tissue sections using color deconvolution and binarized collagen signal analysis in ImageJ software (v1.5)

SUMMARY:
Patients with suspected Lung cancer who underwent contrast-enhanced CT and pathological examinations at Center 1 between January 2011 and January 2020 and Center 2 between September 2017 and Januray 2020 were eligible for inclusion in this study.The Clinical data, preoperative clinical information, laboratory results, CT images and pathological sections were collected. The investigators also collected the disease-free survival and overall survival time. On the Deepwise multi-modal research platform, the images were semi-automatically segmented and PyRadiomics was used to extract the radiomic features. Fibrosis quantification was performed on picrosirius red (PSR)-stained tissue sections using color deconvolution and binarized collagen signal analysis in ImageJ software. The investigators developed RaFIST, a radiomics-based stratification tool, to noninvasively quantify intratumoral fibrosis in non-small cell lung cancer (NSCLC) using contrast-enhanced CT imaging. And it was further tested on the held-out external test cohort. Discrimination was assessed by using the C-index and area under the receiver operating characteristic curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* Solid pulmonary nodule detected on CECT within 3 weeks pre-resection
* No history of previous treatment such as chemotherapy, or radiotherapy

Exclusion Criteria:

* Unavailable pathological sections
* Missing CT images or hard-to-annotate CT images
* Undergone anticancer therapy before CT
* Loss to follow-up
* Concurrent other malignant tumors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Jinling Hospital, China
Sampling Method: Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
DFS (Disease-free survival) | Record from the date of surgery to the date of recurrence or death from any cause, whichever comes first, and assess up to a maximum of 5 years.
  DFS was defined as the duration from the date of primary surgery to the first occurrence of recurrence or death from any cause.

SECONDARY OUTCOMES:
OS (overall survival） | Record from the date of surgery to the date of death from any cause，whichever comes first, and assess up to a maximum of 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No